CLINICAL TRIAL: NCT06380985
Title: Personalized Approach Bias Modification to Reduce Heavy Drinking and Improve Cognitive Control in Veterans With Mild to Moderate Traumatic Brain Injury
Brief Title: Personalized Approach Bias Modification in Heavy Drinking Veterans With Mild to Moderate Traumatic Brain Injury
Acronym: TABM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI resigned from his VA position
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NURA-009-23F; 1I01CX002715-01A1 (Other Grant/Funding Number: Clinical Science Research & Development)
Record Dates: First submitted 2024-04-18; First posted 2024-04-24 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Alcohol Use Disorder; Mild-Moderate Traumatic Brain Injury
Keywords: Cognitive Bias Modification; Alcohol Use Disorder; Brain Injury, Traumatic; Alcohol-Related Disorders; Mental Disorders; Cognitive Training
MeSH Terms: conditions — Alcoholism; Brain Injuries, Traumatic; Alcohol-Related Disorders; Mental Disorders | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: This will be a Phase II double-blind, randomized, sham-controlled clinical trial.
Who Masked: Participant, Investigator
Masking Description: The identity of ApBM and Sham will not be known to investigators or patients. To maintain the blind, the participant and the research coordinator (naïve to ApBM) administering the participant's training will be blind to whether "1" or "2" is ApBM or Sham. The research coordinator will receive the patient assignment from statistical software at time of randomization. The key that determines assignment of ApBM or Sham to condition "1" or "2" will be known by an addiction research program affiliate PI otherwise uninvolved in the current study. They will document this key in a locked electronic file. The study blind will be broken on completion of the study and after the study database has been locked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Personalized VR Alcohol Approach Bias Modification (ApBM) Condition (Experimental): The Personalized VR ApBM will consist of 9 cognitive training sessions, each session lasting approximately 20 minutes completed on separate days over 3 weeks. Each session requires the participant to respond to 240 visual stimuli using a push or pull motion as quickly as possible.
  Interventions: Behavioral: Personalized VR Alcohol Approach Bias Modification (ApBM) Condition
- Sham Condition (Sham Comparator): Sham training will consist of 9 cognitive training sessions, each session lasting approximately 20 minutes completed on separate days over 3 weeks. Each session requires the participant to respond to 240 visual stimuli using a push or pull motion as quickly as possible.
  Interventions: Behavioral: Sham Condition

INTERVENTIONS:
Behavioral: Personalized VR Alcohol Approach Bias Modification (ApBM) Condition — The Personalized VR ApBM will consist of 2D pictures representing alcohol or positive images (e.g., representing family or friends enjoying time together; sports, pets; travel and holidays, etc.) presented in a unique format in VR (e.g., landscape/portrait orientation), which will serve as the cue requiring a stimulus response. Participants are instructed to push the images away from them if they are presented in one format (e.g., landscape) and grab (using lever on VR controller) the images and pull towards themselves in response to a separate format (e.g., portrait pictures) across a virtual table. Each training session starts with 10 practice trials showing neutral objects (containers), followed by 240 training trials (120 alcohol and 120 non-alcohol trials). Training effect is achieved by altering the contingency of push vs. pull by image type (alcohol vs. positive).
  Other Names: ApBM Training
  Arms: Personalized VR Alcohol Approach Bias Modification (ApBM) Condition
Behavioral: Sham Condition — Sham training is identical to ApBM, except the contingency of each orientation (e.g., portrait or landscape) representing a push vs. a pull is altered to diminish training effect.
  Other Names: Sham Training
  Arms: Sham Condition

SUMMARY:
The project will examine the neural associations of alcohol approach-bias and investigate the extent to which a neuroscience-based personalized cognitive training program will remediate alcohol approach-bias and improve recovery outcomes among heavy drinking Veterans with alcohol use disorder (AUD) and a history of mild-moderate traumatic brain injury (mmTBI). Alcohol approach-bias modification (ApBM) is a cognitive training intervention designed to interrupt and modify automatic approach processes in response to alcohol cues. Modification of alcohol approach-bias and reductions in heavy alcohol use can be expected to reduce behaviors of self-harm and violence, increase adherence to medical care, reduce drinking-related medical costs, and promote healthier relationships. The long-term goal is to demonstrate the efficacy of ApBM to promote recovery from AUD in Veterans with chronic mmTBI. The investigators also aim to identify neural mechanisms associated with ApBM and other neurocognitive predictors of successful recovery. The evidence garnered from this study will be useful to inform the development of other behavioral and pharmacological treatments for Veterans with AUD with a history of mmTBI.

DETAILED DESCRIPTION:
This study is the first to test if Alcohol approach-bias modification (ApBM), delivered through virtual reality, as an add-on to outpatient treatment can reduce heavy alcohol use and improve neuro-cognitive outcomes among Veterans with mild to moderate traumatic brain injury (mmTBI) engaged in outpatient treatment for alcohol use disorder (AUD).

This will be a Phase II double-blind, randomized, sham-controlled clinical trial. Approximately 100 heavy drinking Veterans with alcohol use disorder (AUD) and a history of mild to moderate traumatic brain injury (mmTBI) will be randomized into the study to complete a 3-week of either personalized ApBM or sham training (9 training sessions). Immediately following the 3-week training, a post-intervention Week-4 assessment will be administered. The participants will also be re-assessed again at Week 12 as the last study visit.

The aims of the study are as follows:

Aim 1: Establish the efficacy of a personalized alcohol ApBM to promote recovery from AUD among heavy drinking Veterans with a history of mmTBI.

Aim 2: Evaluate alcohol ApBM related change in fMRI cue-induced craving outcomes of treatment response within Default Mode Network.

Aim 3: Assess alcohol approach bias modification-related improvement in cognitive executive functioning domains that typically show deficit in heavy drinking Veterans with mmTBI and replicate preliminary associations between executive function domains and alcohol approach bias.

ELIGIBILITY:
Inclusion Criteria:

* A history of mild-moderate TBI, as defined by American Congress of Rehabilitation Medicine (ACRM), in the chronic, stable phase of recovery (>6 months from injury)
* Heavy drinking defined by NIH/NIAAA criteria (>7 drinks/week for women; >14 drinks/week for men) for at least one week in the last 90 days
* Moderate to severe criteria for current alcohol use disorder (AUD) by DSM-5
* Participants must also be engaged in VA outpatient AUD treatment and express a desire to reduce, stop, or maintain cessation of alcohol use

Exclusion Criteria:

* Unstable clinically significant psychiatric disorders or medical conditions that would create excessive risks, in the clinical judgment of the Principle Investigator
* Current or history of the following:

  * intrinsic cerebral tumors
  * demyelinating and neurodegenerative diseases
  * aneurysm
  * arteriovenous malformations
  * cerebrovascular or peripheral vascular disease
  * severe or penetrating traumatic brain injury
  * documented learning disabilities
  * surgical implantation of neurostimulators or cardiac pacemakers and any other MRI contraindications

    * These conditions/diseases are known to influence the neurocognitive and MR-derived neurobiological measures proposed in this application
* Female participant who is pregnant or actively attempting to conceive (to prevent any unnecessary exposure to high magnetic fields or radiofrequency energy to the unborn child)
* Concurrent participation in another clinical trial on AUD or TBI study
* Requiring acute medical detoxification from alcohol, based on a score of 12 or more on the Clinical Institute Withdrawal Assessment of Alcohol Scale (CIWA-AD)
* Legal mandate to participate in an alcohol treatment program
* Presence of severe TBI or penetrating head trauma
* Starting use of AUD treatment medications (disulfiram, naltrexone, or acamprosate) within the past 4 weeks (must be on AUD treatment for longer than 4 weeks)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Percent of Heavy Drinking Days | 90 days post-randomization
  The primary endpoint is percent of heavy drinking days during the 90 days post-randomization into treatment. A heavy drinking day is defined using NIH/NIAAA criteria, drinking more than 4 drinks a day for men and more than 3 drinks a single day for women.

SECONDARY OUTCOMES:
Cue-induced fMRI BOLD-signal craving activation contrasts | Week 4 - The week following completion of cognitive training.
  BOLD-signal craving activation contrasts (alcohol cues > neutral cues) in amygdala, nucleus accumbens, and posterior cingulate cortex.

OTHER OUTCOMES:
Cognitive flexibility | Week 4 - The week following completion of cognitive training.
  Cognitive flexibility is derived from the Delis-Kaplan Executive Function System (D-KEFS) Trail Making Test Number-Letter Sequencing Condition 4 and Design Fluency Condition 3. Raw scores from these two measures are converted to z-scores based on standard norms. A cognitive flexibility summary score is calculated by averaging the z-scores of the individual constituent measures.

CONTACTS AND LOCATIONS:
Overall Officials: David L Pennington, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA
Locations (1):
- San Francisco VA Medical Center, San Francisco, CA, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No